CLINICAL TRIAL: NCT05483205
Title: Benefit of a Dermocosmetic in Mild to Moderate Adult Acne
Brief Title: Normaderm Phytosolution Global Observational Study
Status: Completed | Type: Observational
Sponsor: Cosmetique Active International (Industry)
Responsible Party: Sponsor
Other Study IDs: NP06072021
Record Dates: First submitted 2022-07-26; First posted 2022-08-02 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-07

CONDITIONS: Acne, Adult
Keywords: acne; observational study; dermocosmetic
MeSH Terms: conditions — Acne, Adult; Acne Vulgaris

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Normaderm Phytosolution Double-Correction Daily Care Moisturizer — Normaderm Phytosolution (NP) was to be applied for up to 90 days once or twice daily, according to the investigator's prescription.
  Other Names: NP

SUMMARY:
The objective of this 3-month observational study was to assess, in 2827 adults, the benefit of NP alone or as adjunctive or maintenance care in mild acne, or as adjunctive care in subjects with moderate acne.

DETAILED DESCRIPTION:
Acne is a chronic inflammatory condition, impacted by exposome factors. A dermocosmetic, Normaderm Phytosolution (NP), was developed to target hyperkeratosis, inflammation, and sebum, while protecting the skin barrier, and to be used either alone or in addition to acne medications. NP is a dermocosmetic specifically developed for acne-prone skin. The lightweight cream is easily absorbed and targets acne pathogenesis thanks to salicylic acid 2% for skin exfoliation, phyco-saccharide 2% for sebum reduction, and vitamin CG as anti-inflammatory ingredient, as well as ingredients that enable regeneration of the disrupted skin barrier, such as Vichy mineralizing water 60%, Bifida ferment lysate 1%, and hyaluronic acid 0.2%.

The study was conducted in accordance with the protocol and the legislative and regulatory provisions in force (after obtaining authorization of the French health authorities and the favorable opinion of the ethics committee).

Qualitative variables were described as numbers and percentages. 95% confidence intervals (CI) were calculated, where required. Quantitative variables were described as number, mean, standard deviation, median, minimum, maximum and number of missing data.

All statistical analyses were performed at a 5% significance using 2-sided tests, except normality, tested at the threshold of 1% (Shapiro-Wilk test).

ELIGIBILITY:
Inclusion Criteria:

Adult men or women (age >18 years old) with mild to moderate acne (GEA scale 1-3).

Exclusion Criteria:

Patients taking isotretinoin. Patients presenting with highly inflammatory acne, grade 4 or 5 on the GEA scale. Patients presenting with nodules.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study took place at 337 sites in 11 countries worlwide. The study population consisted of 2827 patients. Overall, 75.3% were females; mean age was 26.7±8.0 years; 48% of subjects were aged between 18 and 25 years.
Sampling Method: Non-Probability Sample
Enrollment: 2827 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Benefit of NP alone or as adjunctive or maintenance care in mild acne, or as adjunctive care in subjects with moderate acne. | 90-day use
  Change in global acne severity
  using a scale from 0=none to 5 very severe (GEA scale)

SECONDARY OUTCOMES:
Change in seborrhea level | 90-day use
  assessed on a visual analog scale from 0 (absent) to 10 (severe
Change in skin hydration | 90-day use
  assessed on a visual analog scale from 0=no hydration to 10=perfectly hydrated

CONTACTS AND LOCATIONS:
Overall Officials: Delphine Kerob, MD, Study Director — Cosmetique Active International
Locations (11):
- Buenos Aires, Caba, Argentina
- EuroDerma Clinic, Sofia, Bulgaria
- DermaMedEst, Prague, Czechia
- Charite Universitatsklinikum, Berlin, Germany
- Eiffel Esthetics, Budapest, Hungary
- Dermaarte Polanco, Polanco, Mexico
- Polimed, Wroclaw, Poland
- DClinic, Bucharest, Romania
- State Dermatological Clinic #10, Saint Petersburg, Russia
- Amdv s.r.o. kozna amb, Prešov, Slovakia
- Gazi University Medical School, Ankara, Turkey (Türkiye)